CLINICAL TRIAL: NCT01886157
Title: Treatment of Trigger Finger With Steroid Injection Versus Steroid Injection and Splinting: A Randomized Controlled Trial
Brief Title: Treatment of Trigger Finger With Steroid Injection Versus Steroid Injection and Splinting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Philadelphia & South Jersey Hand Center (Other)
Responsible Party: Principal Investigator, Sidney M. Jacoby, Associate Professor, The Philadelphia & South Jersey Hand Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11C.554
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Trigger Finger; Stenosing Tenosynovitis
Keywords: trigger finger; orthotic intervention
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid injection (Active Comparator): Standard corticosteroid injection.
  Interventions: Procedure: Corticosteroid injection
- Corticosteroid Injection and Trigger Splint (Experimental): Corticosteroid Injection + Trigger Splint + Education + Home Exercises
  Interventions: Procedure: Corticosteroid injection + Trigger Splint+ Education and Home exercises

INTERVENTIONS:
Procedure: Corticosteroid injection + Trigger Splint+ Education and Home exercises — Standard corticosteroid injection. Hand based, single digit trigger splint will be applied. Education and instructions about home exercises.
  Arms: Corticosteroid Injection and Trigger Splint
Procedure: Corticosteroid injection — Standard trigger finger corticosteroid injection.
  Arms: Corticosteroid injection

SUMMARY:
Hypothesis: Treatment of trigger finger by corticosteroid injection and splinting is superior to corticosteroid treatment alone.

DETAILED DESCRIPTION:
Stenosing tenosynovitis, or more commonly "trigger finger" is a disease that can severely impact a patient's quality of life. Its incidence is said to be 28 persons per 100,000 annually. The disease is manifested in one or more fingers by finger locking in flexion or extension, leading to pain, discomfort and at times, loss of function. Patients frequently report having to snap their fingers back in position to alleviate symptoms. The pathophysiology relates to thickening of the flexor tendon sheath, which can impair tendon gliding within it.

Although multiple treatment strategies are available, it is not entirely clear which treatment offers the best outcome, especially when the finger has not reached end stage locking. In general, corticosteroid injection into the tendon sheath is offered as the first line of treatment. Splinting alone has also been described as a reliable method treatment. However, Patel and Bassini indicated that steroid injection results in fewer recurrences than splinting alone. Surgery is typically reserved for recurrent triggering, cases refractory to injection, or digits locked in flexion. The effects of steroid injection followed by splinting however have not been reported in a comprehensive fashion. It may be that this form of treatment could result in a synergistic effect, which can offer a treatment modality superior to either injection or splinting alone. The purpose of this research study is to determine whether steroid injection followed by splinting is superior to injection alone.

ELIGIBILITY:
Inclusion Criteria:

* Trigger finger in one or more trigger fingers, in stages 2 to 5 (inclusive)
* Adult patient aged over 18 years.
* No prior treatment (splinting, injection or surgery) to the involved finger OR at least 1 year since last treatment of the involved finger.

Exclusion Criteria:

* Exclude Trigger thumbs because they appear to be respond very favorably or unfavorably to treatment3
* Exclude locked digits because surgery is indicated in these cases
* Pregnant patients
* Prisoners
* Patients with impaired decision-making capacity
* Patients that do not speak English and cannot fill in English language questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Stage of finger triggering | 1, 2, 4-6, and 12 months
  Trigger Finger Stage:
  1. Normal
  2. Painful palpable nodule
  3. Triggering = Clicking = Catching
  4. Locking of finger in flexion or extension unlocked by active finger movement
  5. Locking of finger in flexion or extension unlocked by passive finger movement
  6. Locked finger in flexion or extension (Each stage may be painless or painful)

SECONDARY OUTCOMES:
Failed treatment: surgical intervention required | 1,2, 4-6, 12months
  Failed treatment OR Successful treatment
Patient rated functional outcome | 1, 2, 4-6, 12months
  Quick Disabilities of the Arm, Shoulder and Hand questionnaire Patient Specific Functional Scale
Pain | 1, 2, 4-6, 12 months
  Visual Analog Scale

OTHER OUTCOMES:
Compliance with splint and hand exercises | 1, 2 months
  For patients who are assigned to injection and splint group, home exercise and splint compliance will be assessed by patients maintaining a case log.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Jacoby, MD, Study Director — The Philadelphia and South Jersey Hand Center
Locations (1):
- The Philadelphia and South Jersey Hand Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Ring D, Lozano-Calderon S, Shin R, Bastian P, Mudgal C, Jupiter J. A prospective randomized controlled trial of injection of dexamethasone versus triamcinolone for idiopathic trigger finger. J Hand Surg Am. 2008 Apr;33(4):516-22; discussion 523-4. doi: 10.1016/j.jhsa.2008.01.001. PMID 18406955
- [Result] Strom L. Trigger finger in diabetes. J Med Soc N J. 1977 Nov;74(11):951-4. No abstract available. PMID 269967
- [Result] Colbourn J, Heath N, Manary S, Pacifico D. Effectiveness of splinting for the treatment of trigger finger. J Hand Ther. 2008 Oct-Dec;21(4):336-43. doi: 10.1197/j.jht.2008.05.001. Epub 2008 Aug 22. PMID 19006759
- [Result] Patel MR, Bassini L. Trigger fingers and thumb: when to splint, inject, or operate. J Hand Surg Am. 1992 Jan;17(1):110-3. doi: 10.1016/0363-5023(92)90124-8. PMID 1538090